## Statistical analysis plan

Microsoft Excel was used for data entry and preparation with SPSS version 23 it will be used for statistical analysis. Data will be assessed for normality using Shapiro-Wilk test and groups will be compared using Wilcoxon rank sum test or Student's t-test. A *P*-value <0.05 will be considered statistically significant.